CLINICAL TRIAL: NCT05784545
Title: Highbush Blueberry Supplementation for Osteoarthritis Pain, Intra-articular Inflammation and Post-operative Recovery in Total Knee Replacement Patients
Brief Title: Dietary Supplementation With Blueberry in OA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: U.S. Highbush Blueberry Council (Other); Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRAS Number: 318841
Record Dates: First submitted 2023-03-01; First posted 2023-03-27 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Maltodextrin supplementation
- Blueberry Supplementation (Experimental)
  Interventions: Dietary Supplement: Blueberry powder supplement

INTERVENTIONS:
Dietary Supplement: Blueberry powder supplement — The intervention in this study is 12 weeks of daily blueberry supplementation which is comprised of freeze-dried powdered whole blueberries i.e., blueberries with water removed.
  Arms: Blueberry Supplementation
Dietary Supplement: Maltodextrin supplementation — The intervention in this study is 12 weeks of daily maltodextrin supplement used to mimic the carbohydrate composition of whole blueberries.
  Arms: Placebo

SUMMARY:
Osteoarthritis is a painful long term joint condition that is associated with poor quality of life. There are no treatments to prevent it. Inflammation is one cause of osteoarthritis. This inflammation is complex. It involves many joint tissues, like cartilage and fat. It also involves many proteins that act as inflammatory 'signals'. Safely targeting these proteins with medications has so far proved ineffective. Physiotherapy and weight loss can help osteoarthritis, but there is a need for other approaches. Blueberries are rich in natural chemicals called polyphenols; these have well-established anti-inflammatory effects.

Blueberries and other fruits may improve osteoarthritis symptoms, but the investigators do not know how this improvement happens. It may be that these foods reduce inflammation within the joint tissues. They will investigate this. This will help us to understand 1) how blueberries improve osteoarthritis symptoms and 2) whether dietary supplementation with blueberries could slow down joint damage in osteoarthritis, rather than just improving symptoms. Additionally, high levels of joint inflammation predict poorer recovery from joint replacement surgery. Therefore, blueberry supplementation may hasten this recovery. Fifty eight people scheduled to have a knee replacement for osteoarthritis will receive either six weeks blueberry supplementation or a placebo pre-surgery. Participants will continue the supplementation for six weeks after surgery. First, this study will use tissue samples (cartilage, fat and the joint lining called synovium) obtained during surgery to investigate the effects of pre-operative blueberry supplementation on markers of joint inflammation. Second, this study will assess the ability of dietary supplementation with blueberries to improve the symptoms of osteoarthritis. Finally, this study will investigate the effect of blueberry supplementation on recovery from total knee replacement. Our investigations may provide evidence to support dietary supplementation with blueberries to slow down osteoarthritis progression and to improve recovery from osteoarthritis joint replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participants capable of giving informed consent
* Sex: Male and female
* Age: > 40 years - Those under 40 are more likely to have an undiagnosed secondary cause of osteoarthritis
* BMI: > 18 kg/m2
* Listed to have a total knee replacement for osteoarthritis
* Participants are permitted to participate in other ongoing surgical intervention studies, as long as these are not trials of a dietary supplement or a medication.

Exclusion Criteria:

* Those who have received intravenous or oral immunosuppressant medications in past 2 years
* Those who have had intra-articular steroid injection in 6 months preceding surgery.
* Some secondary causes of osteoarthritis (mechanistic confounders that are likely to influence tissue inflammation measures:
* Known congenital joint disorders
* Other inflammatory arthritis e.g. rheumatoid arthritis
* Avascular necrosis, infectious arthritis
* Paget disease
* Osteopetrosis
* Osteochondritis dissecans
* Hemochromatosis
* Wilson's disease
* Hemoglobinopathy
* Ehlers-Danlos syndrome
* Marfan syndrome
* Acromegaly
* Those typically consuming more than eight 80 g portions (or juice equivalent) of blueberries, blackberries, strawberries, raspberries, blackcurrants, pomegranate or cherries per week
* Those with a known fruit allergy, for which they carry an adrenaline auto-injector or have required anti-histamine, adrenaline, glucocorticoid or beta-agonist treatment.
* Those who cannot adequately understand verbal explanations or written information given in English

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of TNF-ALPHA gene expression in joint tissue (synovium, infrapatellar adipose tissue and cartilage) | In knee at time of surgery (when replaced)
  Inflammatory protein

SECONDARY OUTCOMES:
Concentration of broad panel of Inflammatory and pro-cartilage cytokines samples | Baseline and pre-operatively
  Using multiplex immunoassay including but not limited to at TNFα, IL-6, IL-10 and IL-1β, MIP1α, Galectin 1, Chemerin, Eotaxin, gp130, MCP-1, IL-7, MIP3α, IL-15, Aggrecan, Resistin, Leptin, MIP1β, MMP-1, MMP-3 and MMP-13
Concentration of broad panel of Inflammatory and pro-cartilage degradative gene and protein expression markers | In knee at time of surgery (when replaced)
  Using RTqPCR and immunoblotting including but not limited to TNFα, IL-6, IL1β, IL-8, IL-10, IL-18, IL-7, IL-15, MCP1, LEP, ADIPOQ, NAMPT, RETN, TGFB1, MMP1, MMP2, MMP3, MMP9, MMP13, TIMP1, TIMP2, TIMP3, TIMP4, ADAMTS4, ADAMTS5, , ACAN, COL1A1, COL2A1, COL13A1, COL14A1, COL15A1, DKK1, CCL2, CCL3, CCL4, CCL5, CCL7, CCL8, CCL11, CCL20, CX3CL1, CCR3, CCR2, LGALS1, RARRES2, and IL6ST
Western Ontario and McMaster Universities Arthritis Index Score | Baseline, week 3, week 6, post-surgery, weeks 7, 9 and 12
  Validated questionnaire (0-96 where a higher score is worse)

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Devon University Hospital, Honiton, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No